CLINICAL TRIAL: NCT04819165
Title: Healthcare-associated Infections in Severe COVID-19 Patients Whit Mechanical Ventilation During 2020
Brief Title: Healthcare-associated Infections in Severe COVID-19 During 2020
Acronym: COVIACS
Status: Completed | Type: Observational
Sponsor: Sanatorio Anchorena San Martin (Other)
Responsible Party: Principal Investigator, Matias Accoce, RT, Sanatorio Anchorena San Martin
Other Study IDs: 5/2021
Record Dates: First submitted 2021-03-25; First posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Respiration, Artificial; COVID-19; Health Care Associated Infection
MeSH Terms: conditions — Respiratory Aspiration; COVID-19; Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 patients: Patients with invasive mechanical ventilation admitted to the Intensive Care Unit (UCI) of the Anchorena San Martín Clinic, San Martín, Buenos Aires with confirmed COVID-19 diagnosis (positive polymerase chain reaction in nasopharyngeal swab).
  Interventions: Other: COVID-19
- non COVID-19 patients: Patients with invasive mechanical ventilation admitted to the Intensive Care Unit (UCI) of the Anchorena San Martín Clinic, San Martín, Buenos Aires with negative COVID-19 diagnosis (positive polymerase chain reaction in nasopharyngeal swab).

INTERVENTIONS:
Other: COVID-19 — Impact of covid-19 on infections associated with health care devices.
  Groups: COVID-19 patients

SUMMARY:
In patients who develop ARDS due to SARS-CoV-2 (CARDS), a longer duration of invasive mechanical ventilation (IMV) and ICU stay has been reported compared to ARDS not associated with SARS-CoV-2. Consequently, the days of stay in ICU increase Identifying the risk factors associated with the development of this complication and developing measures aimed at its prevention could have a favorable impact on the clinical course of seriously ill patients.

DETAILED DESCRIPTION:
The rate of catheter-associated bacteremia is 3.78 / 1000 days central venous catheters in polyvalent ICUs.

Some studies suggest that in the context of this pandemic, infections associated with health care have increased, although there are few data referring to Latin America.

The objective of this study is to analyze the incidence of health care associated infections in adult patients on invasive mechanical ventilation with confirmed COVID-19 diagnosis and negative COVID-19 admitted to the Intensive Care Unit of the Anchorena San Martín Clinic, San Martín, Buenos Aires.

ELIGIBILITY:
Inclusion Criteria:

* All patients older than 18 years admitted to the intensive care unit of the Anchorena San Martín Clinic who required invasive mechanical ventilation for more than 24 hours in a period between March 2020 and December 2020 were included in the analysis.

Exclusion Criteria:

* All patients who presented incomplete data in the follow-up sheets were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to ICU who required invasive mechanical ventilation during the COVID-19 pandemic from March to December 2020.
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Incidence of health care associated infections in each group. | March to December 2020

SECONDARY OUTCOMES:
The most frequent pathogens in this population associated with Incidence of health care associated infections. | March to December 2020
Possible factors associated with Incidence of health care associated infections. | March to December 2020
mortality in UCI | March to December 2020
Days of ICU stay | March to December 2020
Days of mechanical ventilation | March to December 2020

CONTACTS AND LOCATIONS:
Overall Officials: matias accoce, Principal Investigator — SAnchorena San Martin
Locations (1):
- Sanatorio Anchorena de San Martin, San Martín, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tufan A, Avanoglu Guler A, Matucci-Cerinic M. COVID-19, immune system response, hyperinflammation and repurposing antirheumatic drugs. Turk J Med Sci. 2020 Apr 21;50(SI-1):620-632. doi: 10.3906/sag-2004-168. PMID 32299202
- [Result] Ripa M, Galli L, Poli A, Oltolini C, Spagnuolo V, Mastrangelo A, Muccini C, Monti G, De Luca G, Landoni G, Dagna L, Clementi M, Rovere Querini P, Ciceri F, Tresoldi M, Lazzarin A, Zangrillo A, Scarpellini P, Castagna A; COVID-BioB study group. Secondary infections in patients hospitalized with COVID-19: incidence and predictive factors. Clin Microbiol Infect. 2021 Mar;27(3):451-457. doi: 10.1016/j.cmi.2020.10.021. Epub 2020 Oct 24. PMID 33223114
- [Result] Bellani G, Laffey JG, Pham T, Fan E, Brochard L, Esteban A, Gattinoni L, van Haren F, Larsson A, McAuley DF, Ranieri M, Rubenfeld G, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Epidemiology, Patterns of Care, and Mortality for Patients With Acute Respiratory Distress Syndrome in Intensive Care Units in 50 Countries. JAMA. 2016 Feb 23;315(8):788-800. doi: 10.1001/jama.2016.0291. PMID 26903337
- [Result] Kalanuria AA, Ziai W, Mirski M. Ventilator-associated pneumonia in the ICU. Crit Care. 2014 Mar 18;18(2):208. doi: 10.1186/cc13775. No abstract available. PMID 25029020
- [Result] Rouze A, Nseir S. Continuous control of tracheal cuff pressure for the prevention of ventilator-associated pneumonia in critically ill patients: where is the evidence? Curr Opin Crit Care. 2013 Oct;19(5):440-7. doi: 10.1097/MCC.0b013e3283636b71. PMID 23856895
- [Result] Duszynska W, Rosenthal VD, Szczesny A, Woznica E, Ulfik K, Ostrowska E, Litwin A, Kubler A. Urinary tract infections in intensive care unit patients - a single-centre, 3-year observational study according to the INICC project. Anaesthesiol Intensive Ther. 2016;48(1):1-6. doi: 10.5603/AIT.2016.0001. PMID 26966105
- [Result] Rosenthal VD, Dwivedy A, Calderon ME, Esen S, Hernandez HT, Abouqal R, Medeiros EA, Espinoza TA, Kanj SS, Gikas A, Barnett AG, Graves N; International Nosocomial Infection Control Consortium (INICC) Members. Time-dependent analysis of length of stay and mortality due to urinary tract infections in ten developing countries: INICC findings. J Infect. 2011 Feb;62(2):136-41. doi: 10.1016/j.jinf.2010.12.004. Epub 2010 Dec 17. PMID 21168440
- [Result] Rouze A, Martin-Loeches I, Povoa P, Makris D, Artigas A, Bouchereau M, Lambiotte F, Metzelard M, Cuchet P, Boulle Geronimi C, Labruyere M, Tamion F, Nyunga M, Luyt CE, Labreuche J, Pouly O, Bardin J, Saade A, Asfar P, Baudel JL, Beurton A, Garot D, Ioannidou I, Kreitmann L, Llitjos JF, Magira E, Megarbane B, Meguerditchian D, Moglia E, Mekontso-Dessap A, Reignier J, Turpin M, Pierre A, Plantefeve G, Vinsonneau C, Floch PE, Weiss N, Ceccato A, Torres A, Duhamel A, Nseir S; coVAPid study Group. Relationship between SARS-CoV-2 infection and the incidence of ventilator-associated lower respiratory tract infections: a European multicenter cohort study. Intensive Care Med. 2021 Feb;47(2):188-198. doi: 10.1007/s00134-020-06323-9. Epub 2021 Jan 3. PMID 33388794